CLINICAL TRIAL: NCT02367963
Title: Evaluation of Comprehensive Lifestyle Peer-group-based Intervention on Cardiovascular Risk Factor, a Randomized Controlled Trial: Fifty-Fifty Program
Brief Title: Peer-group-based Intervention Program
Acronym: Fifty-Fifty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Science, Health and Education, Spain (Other)
Collaborators: Spanish Agency for Consumer, Nutrition and Food Safety (AECOSAN). (Unknown); Nutrition, physical activity and obese prevention Strategy (NAOS) (Unknown); Spanish federation for municipalities and provinces (FEMP). (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SHE-001-FM
Record Dates: First submitted 2015-02-12; First posted 2015-02-20 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases
Keywords: Peer education; Comprehensive health intervention; Lifestyle; Adult; Mid age; Male; Female; Human; Clinical trial; Prevention and control; Cardiovascular Disease; Behavior; Risk Factors; Healthy lifestyle; Healthy people program; Peer-group
MeSH Terms: conditions — Cardiovascular Diseases; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): A Training period and a Peer-group intervention are asigned to this arm. Peer-group intervention is designed to make the subjects participate actively in their healthcare. Through the different activities subjects will begin to successfully make various changes that increase their confidence in the ability to manage risk factors and problems arising from unhealthy habits. Along the twelve sessions (60-90 minutes) subjects propose assumable health goals; learn to manage their emotions, to resolve problems, to control their diet, to increase their physical activity, to control their state of mind and how the acquisition or not of healthy habits influences their relationships.
  Interventions: Behavioral: Training period; Behavioral: Peer-group
- Control (Other): A Training period intervention is asigned to this arm. Once the workshops have been carried out, the control group will be provided with written and visual documentation of risk factors and overall health habits. The members of this group will have access to the study website, where they will be able to find information on risk factors and health habits and links to the same websites related to health as the intervention group.
  They won't participate in the sessions of peer education group dynamics for a period of 12 months.
  Interventions: Behavioral: Training period

INTERVENTIONS:
Behavioral: Training period — Six workshops in which education on health habits and encouragement to reduce risk factors was promoted. Workshops addressed rigorous, accurate and effective technical information but were tailored to general public to ensure that subjects became aware of the importance of change in their overall health. Workshops led by experts dealt with the following relevant subjects: Motivation to Change; Physical Activity, Healthy Diet, Smoking Cessation; Stress Management and Self-control of Blood Pressure.
Behavioral: Peer-group — The ultimate goal is to reinforce the self-accountability in the subjects and nurture their self-care. It is designed to make the subjects participate actively in their healthcare. Through the different activities subjects will begin to successfully make various changes that increase their confidence in the ability to manage risk factors and problems arising from unhealthy habits. Along the twelve sessions (60-90 minutes) subjects propose assumable health goals; learn to manage their emotions, to resolve problems, to control their diet, to increase their physical activity, to control their state of mind and how the acquisition or not of healthy habits influences their relationships.
  Arms: Intervention

SUMMARY:
Cardiovascular disease is the leading cause of death in Spain and worldwide. Interventions targeting dietary patterns, weight reduction and new physical activity habits often result in impressive rates of initial behavior changes, but frequently these are not translated into long term maintenance. We hypothesize that a peer-group intervention, addressing multiple facets of cardiovascular disease risk factor can be successfully implemented improving the adherence of participants to healthy habits.

A multicenter, randomized control trial scheme was adopted. A peer-group based intervention approach in which community members support each other to promote health-enhancing changes was chosen. Around 600 participants from 7 Spanish municipalities received a 12h initial training and were randomly allocated to intervention or control groups for a 12-month peer intervention. Baseline measurements took place before and after the initial training. Follow-up measurements will be taken at the end of the intervention and 1 and 2 years after the end of the study. The primary outcome is the improvement in a newly defined score combining 5 individual variables. Secondary outcomes are 1, 2 and 3 years variations in anthropometric parameters and/or healthy behaviors.

The project seeks the empowerment of subjects from 25 to 50 years of age to improve their overall health habits and self-control of risk factor through peer education. The initiative is being developed in cooperation with the Spanish Agency for Consumer Affairs, Food Safety and Nutrition (AECOSAN). This study will allow the economic and feasibility evaluation of the intervention, which will enable policy makers to consider its potential wider implementation for a real community-based intervention.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of death in Spain and worldwide. Obesity, smoking, physical inactivity and high blood pressure act as major risk factors. Although these major risk factors cannot be necessarily eliminated developing healthy habits and behaviors can reduce the possibilities of heart attacks.

The hypothesis of the project focuses on the thought that if adults are trained, among peers, and are provided with new knowledge, skills and attitudes on a healthy lifestyle their cardiovascular health and self-control of risk factors will improve.

The main objective of this comprehensive intervention is to explore the evolution of multiple cardiovascular diseases, risk factor including blood pressure, body mass index (BMI) and waist circumference.

The project is a pilot study for a community intervention, multicenter, randomized, controlled and longitudinal in nature for a period of 15 months, lasting the intervention 12 months. Besides, the project entails a follow-up after 2 year.

The overall approach of the study is as follows:

1. Recruitment: For participant recruitment, town council representatives were contacted by the management team and a strategy was designed for the publicity of the project among the town population. A representative from the town council designed as the coordinator for the local municipality works in close collaboration with the project team. Once potential subjects were identified, a recruiting meeting was held in which the overall project objective is presented.
2. Inclusion: Volunteers that expressed their interest in participating in the program were examined for inclusion criteria. Eligible participants are aged 25-50 and present at least one of the following cardiovascular risk factor and/or lifestyle-related risk factor: hypertension (≥140/90 or ≤140/90 under treatment), overweight or obesity (BMI ≥25), smoking (Smoker), or physical inactivity (≤150min/week).

   Those acceptable were included and registered at the program's website. A more detailed and in-depth explanation of the program was then given to the selected subjects in a second meeting. Afterwards subjects were invited to sign the informed consent and to acknowledge the program's objectives.
3. Baseline Assessment (A1): the physical annotations of the subjects are carried out. Variables such weight, height, waist perimeter and blood pressure and the calculation of the BMI are measured. Additionally information related to eating habits, smoking, physical activity, quality of life, and socio-demographic data is collected using the online questionnaire.

   All participants followed a training period consisting on six workshops in which education on health habits and encouragement to reduce risk factors was promoted. Workshops addressed rigorous, accurate and effective technical information but were tailored to general public to ensure that subjects became aware of the importance of change in their overall health.
4. Assessment 2 (A2): after two months and the workshops' completion, at which contact details are reassured and the non-occurrence of any of the exclusion criteria is confirmed, repeated measures of body weight, waist perimeter, blood pressure and surveyed habits are assessed.

   After the training period, those who did not attend the workshops and the second assessment were excluded from the study. The remaining accepted participants were then randomized to either control or interventional groups using the sex as stratification factor to ensure that the groups were balanced by sex.

   To promote reduction of cardiovascular diseases risk, the Fifty-Fifty program uses evidenced-based recommendations for cardiovascular diseases prevention.

   The intervention is designed to promote the active participation of subjects in their own healthcare. The ultimate goal of the program, and specifically that of the intervention, is to reinforce the self-accountability of the subjects and nurture their self-care. The approach for health promotion is the peer education, in which community members support themselves promoting health-enhancing changes among peers.

   The participants are randomly assigned to subgroups for the intervention. The intervention is initiated by health, education and psychology professionals who help recruiting two volunteers from each subgroup to serve as peer educators or leaders.

   For selecting the leaders, each subgroup goes through a preset group-dynamics education directed by an expert psychologist, for assessing group members for leadership, availability for the role and clear understanding of the intervention. For preparing the chosen leaders as peer educators, they are trained in a 3-hour session on relevant health and health-promotion information, leadership and communication skills.

   Twelve peer-group meetings will be held on a monthly basis and each meeting will last for 60-90 minutes. The activities involved in the group dynamics will include, at their own choice, group discussions, role-playing, brainstorming, relaxation techniques, menu design, joint sportive activities, and others. These activities will directly stimulate the incorporation of healthy habits by participants and will enhance their confidence in their ability to manage risk factor and problems arising from healthy habits. At each meeting, participants will address emotion management, problem resolution, relapse prevention, diet control and physical activity engagement. Through these reflections participants will propose affordable goals that will improve their life style.

   As a fundamental instrument for increasing awareness on healthy habits and self-control of cardiovascular diseases risk factor, participants are provided with a health handbook to register their health parameters and will record their immediate goals at each group meeting. Progress and new goals will be discussed in the context of the whole group.

   An important aspect of the program is empowering individuals for the self- monitoring of blood pressure. Blood pressure is a main target of the intervention and is directly related to most healthy habits specifically targeted in this study. Automated blood pressure measuring devices will be donated to participants for their own use and appropriate training on the use of the devices is provided. Through this action participants will then directly control a fundamental aspect of their cardiovascular diseases risk. Due to its special relevance, a specific blood pressure registry card will be provided for the follow up of participants blood pressure during the whole study.

   In addition, for increasing the awareness on their situation and evolution, participants receive a copy of the score card in which the objective evaluation of their cardiovascular diseases risk factor is determined.
5. Assessment at the end of the 12-month intervention (A3): this assessment is carried out upon the 15-month duration of the study. Again contact details are reconfirmed and repeated measures such as body weight, waist perimeter, blood pressure and surveyed habits are collected.
6. Assessment (A4): this assessment is carried out one year after the intervention.
7. Final assessment (A5): this assessment is carried out two year after the intervention.

Data obtained:

1. Anthropometric data: blood pressure, weight, height and waist circumference.
2. Healthy habits are collected by standardized questionnaires
3. Self-controlled blood pressure (BP) data are also obtained in the intervention group. A frequency of self-measures (2 per day -2 days per week - 2 weeks per month) is intended and will generate a total of 96 measures.

Data registry: the SHE Foundation owns the project database. It is registered with the Spanish Agency for Data Protection under the name of the Fifty-Fifty Program.

A responsible for the database coordinates the management of the all data arising from the study and monitors the quality control.

Personal data will be introduced by each of the subjects at the time of registration. Once this data is included in the web application and a subject is selected by the research team, the computer system will send a code and password to each of them ensuring the anonymity of the assessment data arising from the study. If a subject has any troubles accessing the database information the responsible is there to facilitate his/her accessibility.

The data from the physical assessment-weight, height, waist perimeter, blood pressure-will be collected by those trained for the purpose, and will be uploaded into the system; again, ensuring the highest standards of confidentiality and security. The data collected will be verified by the responsible for the database.

An essential part of the study is data anonymization to comply with current regulations and legislation. At the moment that the subject enters the study, the system will assign him/her an identification (ID) number that will be unique and exclusive to that subject. Each subject's visit will be recorded by a code associated with his/her ID number. This will guarantee that the information appearing in a list is anonymous and cannot be credited to any specific individual.

The processing of the data will conform to the provisions of the Organic Law 15/1999, December, 13, regarding the protection of personal data. Access to the subject information is restricted to a very limited part of the staff involved in the study, but always maintaining absolute confidentiality thereof and complying with current legislation therefrom.

The website database will contain all the study information including data from different explorations, survey information and data on the progress of the scores of both the initial and longitudinal phases of the study. The database will be centralized and will be unique to avoid redundancies and inconsistencies. The information contained in the database will have followed a rigorous quality control.

Ethical concerns: Informed written consent for participation is required from the participants to become part of the study. The written consent specifies the purpose of the study and the intervention, test and measures that are going to be taken. Participants are also notified that withdrawal at any time is immediate and without any consequences. We assure the confidentiality of all the data submitted and measures taken from the participants. The information collected is treated according to the organic law 215/1999 for the protection of personal data. Ethical approval was received from a committee of reference.

Statistical analysis: The percentage of individuals in the intervention and control groups who substantially improve their health habits will be estimated. Based on power calculations, a difference of at least 15% between the intervention and control groups will be detected. Assuming and approximate 10% loss to follow-up and/or refusal to participate, the minimum number of subjects needed in each group to detect this change is 250 participants.

A descriptive analysis of the population based on selected variables will be carried out at baseline and follow up. The prevalence of overweight, obesity, hypertension, smoking, physical inactivity and adherence to Mediterranean diet in both groups by sex and age (from 25 to 34 and 35 to 50 years) in each of the 3 assessments will be calculated. Total Fuster-BEWAT score (combination of 5 variables: blood pressure, exercise, weight, alimentation and tobacco) values will be computed. The percentages of subjects who have increased their total score from the beginning of the program to its completion will be determined. A comparison test of proportions for independent samples will be used to assess whether significant changes have occurred in the total score and in the various dimensions of the score, assuming as statistical significance the value of p<0.05. Student's t-test will be used to assess whether the average score at the end of the program is significantly different in both intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must sign the informed consent and acknowledge the program's objectives.
* Subjects must be born between 1963 and 1988 both inclusive.
* Subjects must at least present one of the following characteristics:

  * To be overweight or obese: BMI ≥ 25 kg/m2
  * To be physically inactive: carry out less than 150 minutes of exercise a week for periods not less than 10 minutes
  * To be a smoker
  * To have high blood pressure

Exclusion criteria:

* To be unable to meet any of the inclusion criteria
* To have been pregnant in January 2013 or to get pregnant during the program
* To have a history of any of the chronic diseases given below:

  * Cardiovascular disease
  * Cerebrovascular disease
  * Diabetes mellitus
  * Other metabolic or endocrine diseases requiring continuous treatment
  * Pathological oncology
  * Inflammatory bowel disease
  * Any other disease of chronic nature requiring continuous treatment with immunosuppressive drugs or corticosteroid therapy
  * Other reasons and any other disease after the baseline assessment

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 543 (Actual)
Dates: Start 2013-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The improvement in a newly defined score combining 5 individual variables: the Fuster-BEWAT score | 1,2 and 3 year follow-up after the intervention.
  The primary outcome measure is the mean change in the overall Fuster-BEWAT score, which assimilates scores related to Blood pressure, Exercise, Weight, Alimentation and Tobacco. The primary outcome is whether individuals belonging to a lifestyle intervention program (intervention group) demonstrate an improvement of health related behaviors and biological parameters compared to the self-management approach (control group).

SECONDARY OUTCOMES:
The mean changes in the individual components of the Fuster-BEWAT score and the mean changes in systolic and diastolic blood pressure levels and Body Mass Index and in the habit parameters evaluated using validated questionnaires. | 2 and 3 years
  Anthropometric data of the subjects such weight, height, waist circumference and blood pressure are measured.
  Information related to eating habits, smoking, physical activity, quality of life, and socio-demographic data is collected using questionnaires:
  * The standardized International Phisical Activity Questionnaire (IPAQ).
  * The shortened Fagerström dependency and the Richmond questionnaires regarding smoking.
  * The "Prevención con dieta mediterránea" (PREDIMED) validated 14-item screening tool for measuring adherence to the Mediterranean diet.
  * A reduced version of SF36 (health survey to measure the overall health) questionnaire for measuring the quality of life.
  * In addition, all participants are asked to provide socio-demographic and report on readiness to change or improving healthy behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Valentín Fuster, MD, PhD, Study Chair — Chairman of the Foundation for Science for Health and Education; Emilia Gómez Pardo, PhD, Principal Investigator — Scientific Director Foundation for Science for Health and Education
Locations (1):
- Foundation for Science, Health & Education, Madrid, Spain, Spain

REFERENCES:
- [Derived] Fernandez-Alvira JM, Fernandez-Jimenez R, de Miguel M, Santos-Beneit G, Bodega P, Hill CA, Carral V, Rodriguez C, Carvajal I, Orrit X, de Cos-Gandoy A, Dal Re M, Robledo T, Fuster V. The challenge of sustainability: Long-term results from the Fifty-Fifty peer group-based intervention in cardiovascular risk factors. Am Heart J. 2021 Oct;240:81-88. doi: 10.1016/j.ahj.2021.06.006. Epub 2021 Jun 18. PMID 34147462
- [Derived] Gomez-Pardo E, Fernandez-Alvira JM, Vilanova M, Haro D, Martinez R, Carvajal I, Carral V, Rodriguez C, de Miguel M, Bodega P, Santos-Beneit G, Penalvo JL, Marina I, Perez-Farinos N, Dal Re M, Villar C, Robledo T, Vedanthan R, Bansilal S, Fuster V. A Comprehensive Lifestyle Peer Group-Based Intervention on Cardiovascular Risk Factors: The Randomized Controlled Fifty-Fifty Program. J Am Coll Cardiol. 2016 Feb 9;67(5):476-85. doi: 10.1016/j.jacc.2015.10.033. Epub 2015 Nov 9. PMID 26562047